CLINICAL TRIAL: NCT01823341
Title: Outpatient Reduction of Nocturnal Hypoglycemia by Using Predictive Algorithms and Pump Suspension in Children
Acronym: PSO4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PSO4; 5R01DK085591 (NIH)
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Results first posted 2015-08-24 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Hypoglycemia; Continuous Glucose Monitoring; Pump Suspension
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pump suspension algorithm (Active Comparator): The pump suspension algorithm will be running actively on the study laptop during the night and suspend the pump if the algorithm predicts hypoglycemia.
  Interventions: Device: Pump suspension algorithm
- Standard of Care (No Intervention): The control algorithm will run passively and not suspend the patient's pump.

INTERVENTIONS:
Device: Pump suspension algorithm — The study laptop will communicate to the pump causing a suspension based on output from the algorithm which predicts hypoglycemia.
  Arms: Pump suspension algorithm

SUMMARY:
The purpose of this study is to see whether low blood sugar at night can be reduced by using a system that turns off the insulin pump automatically. The study system includes a continuous glucose monitor (CGM) and an insulin pump. The CGM and pump work with a regular laptop computer. A The system works by (1) measuring the glucose levels under the skin with the CGM, (2) using a computer program on the laptop to predict whether a low blood sugar is likely to occur, and (3) turning off the insulin pump when the computer program predicts that a low blood sugar will occur.

We have tested the system in the home environment in individuals with type 1 diabetes age 15 years and older. We have found an indication that the system can decrease the frequency of hypoglycemia. We have not had any serious cases of high blood sugars or other problems. We are now ready to further test the system in the home environment in a younger age group to learn more about its ability to reduce overnight low blood sugar risk.

This study has several phases and will take about 3 months for a patient to complete.

* First, the patient will use the CGM and pump at home for up to 15 days with the help of a parent/guardian. This is done to determine if the patient meets our study criteria to proceed with the next phase of the study.
* If the patient is eligible to continue in the study, the patient will need to use the full study system for at least 5 nights at home with the help of a parent/guardian. This is done to make sure the patient and parent/guardian are able to use the system correctly. The patient may participate in starting and stopping the system at home, but the parent/guardian is responsible for making sure it is used as instructed.
* After that, the patient will be asked to use the study system each night for an additional 6 to 8 weeks. The parent/guardian will remain responsible for making sure the system is used as instructed.

The study will include about 90 individuals with type 1 diabetes at 3 clinical centers in the United States and Canada. First a study of children 8 to less than 15 years old will be done. Then, a study of children 3 to less than 8 years old will be conducted.

DETAILED DESCRIPTION:
Patients who are eligible for the clinical trial initially will use a Veo insulin pump and Enlite sensor at home to verify that the patient is able to use the continuous glucose monitor (CGM) and insert sensors and is eligible to continue in the study. A parent or guardian of the child subject will oversee the actions of the subject and be responsible for the patient's overall participation during the proposed study, including operation of the investigational device system.

The first 10 patients 8 to <15 years of age will participate in an Algorithm Assessment Phase of approximately 10 nights of active system use each (for a nominal total of 100 nights of use) to determine if any adjustments to the algorithm parameters are needed and if it is safe to advance to a randomized clinical trial phase with these subjects. If adjustments are needed, the Algorithm Assessment Phase will be repeated, using the same 10 patients if possible. Once the randomized clinical trial phase begins for patients 8 to <15 years of age, approximately 200 nights of randomized system use will be collected and assessed for safety before any patients 3 to <8 years of age may be enrolled in the study. When enrollment does begin for patients 3 to <8 years of age, a second Algorithm Assessment Phase will be conducted with the first 10 patients in that younger age group using the same approach described above for the older subjects. Once the randomized clinical trial phase begins for patients 3 to <8 years of age, a final Data Safety Monitoring Board safety assessment will be performed after approximately the first 200 nights of randomized system use.

Patients who enroll in the study after the completion of the Algorithm Assessment Phase for their age group will use the closed-loop system at home for at least 5 days to demonstrate their ability to use the system and submit study data to the Coordinating Center.

Patients who successfully demonstrate their ability to use the system at home as described above will be eligible for the randomized trial phase. This phase consists of use of the full system as an outpatient for approximately 42 nights:

* Each night the blood glucose (BG) level will be checked with the BG meter and used to perform a calibration of the CGM. This calibration must occur no more than 90 minutes prior to activation of the system. NOTE: Subjects will be instructed to calibrate the CGM per manufacturer guidelines.
* Then the system will be activated, linking the CGM and insulin pump to the computer at the bedside.
* A randomization schedule on the laptop will be used to determine whether the 'pump shut off' application will be active that night or not.
* Patients will be blinded as to whether the pump shut off is active when a session is initiated each night.
* There will not be an alarm if the pump shuts off. The CGM alarm will be set to 60 mg/dL (3.3 mmol/L). When a CGM alarm occurs, the subject will be asked to measure the blood glucose with a BG meter, if he/she is aware of the alarm.
* Patients will be asked to check blood ketones with the study ketone meter if the subject has a fingerstick BG ≥250 mg/dL (13.9 mmol/L).
* Patients will be asked to check blood glucose with the study BG meter, blood ketones with the study ketone meter, and urine ketones with a ketone strip each morning prior to breakfast and enter the results using the controller software interface. The patient will be instructed to contact the study physician if the blood glucose or ketone readings are out of an expected range.
* Patients will be asked to record all overnight carbohydrate intake using the controller software interface.
* Patients will be asked to perform periodic CGM data uploads using the controller software interface.

Upon completion of the study, patients as well as study clinicians will be asked to complete a human factors usability questionnaire regarding use of the study system.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year and an insulin infusion pump for at least 6 months
* Age 3 to <15 years
* HbA1c <=8.5%
* Availability of internet access for periodic upload of study data

Exclusion Criteria:

* Diabetic ketoacidosis in the past 3 months
* Hypoglycemic seizure or loss of consciousness in past 6 months
* History of seizure disorder (except for hypoglycemic seizures)
* Cystic fibrosis
* Current use of oral/inhaled glucocorticoids, beta-blockers or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
* History of ongoing renal disease (other than microalbuminuria), or liver disease (Creatinine is > 1.5 mg/dL (132 µmol/L))
* Medical or psychiatric condition that in the judgment of the investigator might interfere with the completion of the protocol such as:

  * Inpatient psychiatric treatment in the past 6 months
  * Uncontrolled adrenal disorder
  * Abuse of alcohol
* Pregnancy
* Liver disease as defined by an Alanine Aminotransferase Test (ALT) greater than 3 times the upper limit of normal

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy W Beck, MD, PhD, Principal Investigator — Jaeb Center for Health Research; Bruce A Buckingham, MD, Study Chair — Stanford University; John Lum, MS, Study Director — Jaeb Center for Health Research
Locations (3):
- United States (2):
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
- St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Result] Buckingham BA, Raghinaru D, Cameron F, Bequette BW, Chase HP, Maahs DM, Slover R, Wadwa RP, Wilson DM, Ly T, Aye T, Hramiak I, Clarson C, Stein R, Gallego PH, Lum J, Sibayan J, Kollman C, Beck RW; In Home Closed Loop Study Group. Predictive Low-Glucose Insulin Suspension Reduces Duration of Nocturnal Hypoglycemia in Children Without Increasing Ketosis. Diabetes Care. 2015 Jul;38(7):1197-204. doi: 10.2337/dc14-3053. Epub 2015 Jun 6. PMID 26049549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at Stanford University (Stanford, CA), the Barbara Davis Center (Denver, CO), and Children's Hospital, London Health Sciences Centre (London, ON). A total of 53 subjects 11-14 years old and 44 subjects 4-10 years old were enrolled. Forty-five of the 11-14 year old subjects and 37 of the 4-10 year old subjects completed.
Pre-assignment Details: After the run-in phase, a 42-night randomized trial was conducted in which each night was randomly assigned to have either predictive low glucose suspend system active (intervention) or inactive (control) with half of the nights being intervention and half control nights.
Groups:
- Randomized Nights- Treatment or Control: Each study night will be randomized to have either Predictive Low Glucose Suspend or to be inactive (control). On nights randomized to the intervention treatment, the study laptop will be running actively during the night and suspending the patient's pump if the algorithm predicts hypoglycemia based on the patient's continuous glucose sensor trend. (Pump suspension : The study laptop will communicate to the pump causing suspension based on output from the algorithm which predicts hypoglycemia based on the continuous glucose sensor trend.) On control nights, the algorithm will run passively and not recommend suspensions or resumption to the patient's pump.
Period: Overall Study
Arm/Group | Randomized Nights- Treatment or Control
Started | 97
Completed | 82
Not Completed | 15
Not completed — Failed run-in | 7
Not completed — Withdrawal by Subject | 7
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: 45 Subjects age 11-14 years and 37 subjects age 4-10 years
Arm/Group | Randomized Nights- Treatment or Control
Number analyzed (Participants) | 82
Age, Customized [Median (Inter-Quartile Range); unit: years]
  11-14 Year olds | 13 [11 to 13]
  4-10 Year olds | 8 [6 to 9]
Sex/Gender, Customized [Number; unit: participants]
  Male Participants 11-14 year old age group | 25
  Female Participants 11-14 year old age group | 20
  Male Participants 4-10 year old age group | 17
  Female Participants 4-10 year old age group | 20
Race/Ethnicity, Customized [Number; unit: participants]
  White non-Hispanic Participants 11-14 years old | 43
  Hispanic Participants 11-14 years old | 1
  Asian Participants 11-14 years old | 1
  White non-Hispanic Participants 4-10 years old | 35
  Hispanic Participants 4-10 years old | 2
  Asian Participants 4-10 years old | 0
Diabetes Duration [Median (Inter-Quartile Range); unit: years]
  Participants 11-14 years old | 6 [3 to 9]
  Participants 4-10 years old | 3 [2 to 5]
Body-mass index percentile (BMI) [Median (Inter-Quartile Range); unit: BMI Percentile] — Body-mass index percentiles adjusted for age and gender were computed using the 2000 CDC population growth chart data (Kuczmarski RJ, Ogden CL, Grummer-Strawn LM, et al. CDC growth charts: United States. Adv Data 2000:1-27).
  BMI Percentile
    Participants 11-14 years old | 69 [44 to 82]
    Participants 4-10 years old | 69 [51 to 82]
HbA1c (%) [Median (Inter-Quartile Range); unit: Percent]
  Participants 11-14 years old | 7.7 [7.3 to 8.2]
  Participants 4-10 years old | 7.8 [7.5 to 8.0]
HbA1c (mmol/mol) [Median (Inter-Quartile Range); unit: mmol/mol]
  Participants 11-14 years old | 61 [56 to 66]
  Participants 3-10 years old | 62 [58 to 64]
Daily insulin dose (U/kg/day) [Median (Inter-Quartile Range); unit: U/kg/day]
  Participants 11-14 years old | 0.83 [0.72 to 0.96]
  Participants 4-10 years old | 0.76 [0.69 to 0.86]

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Time Spent in Hypoglycemia (<70 mg/dl, 3.9 mmol/L) Overnight on Intervention Nights Versus Control Nights, Normalized to an 8-hour Period.
Description: Each night is categorized as to whether hypoglycemia occurred. Hypoglycemia is defined as the occurrence of one or more CGM glucose values ≤70 mg/dL (3.9 mmol/L). The time period for outcome assessment each night will be from the time the system is activated in the evening until the time it is deactivated in the morning. The percentage of hypoglycemic nights (CGM glucose value ≤70 mg/dL (3.9 mmol/L)) will be tabulated separately with versus without the closed-loop control system in use. We considered nights with at least 4 hours of sensor glucose data as a "valid" night toward the 42 night overall goal and thus our final analyses had a slightly higher number of nights than expected.
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use.
Population: One participant in the 4-10 year old age group with 5 intervention nights and 5 control nights was excluded for <80h of CGM glucose data. We considered nights with at least 4 hours of sensor glucose data as a "valid" night toward the 42 night overall goal and thus our final analyses had a slightly higher number of nights than expected.
Measure: Median (Inter-Quartile Range); unit: percentage of time
Units Other Than Participants: Number of Nights Analyzed
Groups:
- Pump Suspension Algorithm (Participants 11-14 Years); Pump Suspension Algorithm (Participants 4-10 Years): The study laptop will be running actively during the night and suspending the patient's pump if the algorithm predicts hypoglycemia based on the patient's continuous glucose sensor trend.
  Pump suspension: The study laptop will communicate to the pump causing a suspension based on output from the algorithm which predicts hypoglycemia based on the continuous glucose sensor trend.
- Standard of Care (Participants 11-14 Years); Standard of Care (Participants 4-10 Years): The control algorithm will run passively and not recommend control the patient's pump.
Arm/Group | Pump Suspension Algorithm (Participants 11-14 Years) | Standard of Care (Participants 11-14 Years) | Pump Suspension Algorithm (Participants 4-10 Years) | Standard of Care (Participants 4-10 Years)
Number analyzed (Participants) | 45 | 45 | 36 | 36
Number analyzed (Number of Nights Analyzed) | 955 | 941 | 769 | 755
percentage of time | 4.6 [2.9 to 7.3] | 10.1 [5.9 to 13.8] | 3.1 [1.6 to 5.0] | 6.2 [3.0 to 7.6]
Statistical Analysis 1: Comparison: Pump Suspension Algorithm (Participants 11-14 Years) vs Standard of Care (Participants 11-14 Years) vs Pump Suspension Algorithm (Participants 4-10 Years) vs Standard of Care (Participants 4-10 Years); Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Percentage of Nights With 1 or More Sensor Glucose Values <70 mg/dL (<3.9 mmol/L)
Description: Please note we considered nights with at least 4 hours of sensor glucose data as a "valid" night toward the 42 night overall goal and thus our final analyses had a slightly higher number of nights than expected.
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use.
Population: One participant in the 4-10 year old group with 5 intervention nights and 5 control nights was excluded for <80h of CGM glucose data. We considered nights with at least 4 hours of sensor glucose data as a "valid" night toward the 42 night overall goal an thus our final analyses had a slightly higher number of nights than expected.
Measure: Number; unit: percentage of nights
Units Other Than Participants: Nights Analyzed
Arm/Group | Pump Suspension Algorithm (Participants 11-14 Years) | Standard of Care (Participants 11-14 Years) | Pump Suspension Algorithm (Participants 4-10 Years) | Standard of Care (Participants 4-10 Years)
Number analyzed (Participants) | 45 | 45 | 36 | 36
Number analyzed (Nights Analyzed) | 955 | 941 | 769 | 755
percentage of nights | 34 | 39 | 28 | 33
Statistical Analysis 1: Comparison: Pump Suspension Algorithm (Participants 11-14 Years) vs Standard of Care (Participants 11-14 Years); Test type: Superiority or Other; p = 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Pump Suspension Algorithm (Participants 4-10 Years) vs Standard of Care (Participants 4-10 Years); Test type: Superiority or Other; p = 0.04, t-test, 2 sided

3. Secondary Outcome: Percentage of Nights With 1 or More Sensor Glucose Values <50 mg/dL (<2.8 mmol/L)
Description: as for outcome 2
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Population: as for outcome 2
Measure: Number; unit: percentage of nights
Units Other Than Participants: Nights analyzed
Arm/Group | Pump Suspension Algorithm (Participants 11-14 Years) | Standard of Care (Participants 11-14 Years) | Pump Suspension Algorithm (Participants 4-10 Years) | Standard of Care (Participants 4-10 Years)
Number analyzed (Participants) | 45 | 45 | 36 | 36
Number analyzed (Nights analyzed) | 955 | 941 | 769 | 755
percentage of nights | 12 | 17 | 10 | 14
Statistical Analysis 1: Comparison: Pump Suspension Algorithm (Participants 11-14 Years) vs Standard of Care (Participants 11-14 Years); Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Pump Suspension Algorithm (Participants 4-10 Years) vs Standard of Care (Participants 4-10 Years); Test type: Superiority or Other; p = 0.005, t-test, 2 sided

4. Secondary Outcome: Mean Sensor Glucose Overnight
Description: as for outcome 2
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Population: One participant in the 4-10 year old age group with 5 intervention nights and 5 control nights was excluded for <80h of CGM glucose data. We considered nights with at least 4 hours of sensor glucose data as a "valid" night toward the 42 night overall goal an thus our final analyses had a slightly higher number of nights than expected.
Measure: Mean (Standard Deviation); unit: mg/dL
Units Other Than Participants: Nights Analyzed
Arm/Group | Pump Suspension Algorithm (Participants 11-14 Years) | Standard of Care (Participants 11-14 Years) | Pump Suspension Algorithm (Participants 4-10 Years) | Standard of Care (Participants 4-10 Years)
Number analyzed (Participants) | 45 | 45 | 36 | 36
Number analyzed (Nights Analyzed) | 955 | 941 | 769 | 755
mg/dL | 152 (19) | 144 (18) | 160 (16) | 153 (14)
Statistical Analysis 1: Comparison: Pump Suspension Algorithm (Participants 11-14 Years) vs Standard of Care (Participants 11-14 Years); Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Pump Suspension Algorithm (Participants 4-10 Years) vs Standard of Care (Participants 4-10 Years); Test type: Superiority or Other; p = 0.004, t-test, 2 sided

5. Secondary Outcome: Percentage of Time Overnight Sensor Glucose Values 71 to 180 mg/dL (3.9 to 10.0 mmol/L), Normalized to an 8-hour Period.
Description: as for outcome 2
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of time
Units Other Than Participants: Nights analyzed
Arm/Group | Pump Suspension Algorithm (Participants 11-14 Years) | Standard of Care (Participants 11-14 Years) | Pump Suspension Algorithm (Participants 4-10 Years) | Standard of Care (Participants 4-10 Years)
Number analyzed (Participants) | 45 | 45 | 36 | 36
Number analyzed (Nights analyzed) | 955 | 941 | 769 | 755
percentage of time | 66 (10) | 64 (10) | 63 (11) | 63 (10)
Statistical Analysis 1: Comparison: Pump Suspension Algorithm (Participants 11-14 Years) vs Standard of Care (Participants 11-14 Years); Test type: Superiority or Other; p = 0.10, t-test, 2 sided
Statistical Analysis 2: Comparison: Pump Suspension Algorithm (Participants 4-10 Years) vs Standard of Care (Participants 4-10 Years); Test type: Superiority or Other; p = 0.50, t-test, 2 sided

6. Secondary Outcome: Percentage of Overnight Time Spent With CGM Value >250 mg/dL (13.9 mmol/L), Normalized to an 8-hour Period.
Description: as for outcome 2
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percentage of time
Units Other Than Participants: Nights Analyzed
Arm/Group | Pump Suspension Algorithm (Participants 11-14 Years) | Standard of Care (Participants 11-14 Years) | Pump Suspension Algorithm (Participants 4-10 Years) | Standard of Care (Participants 4-10 Years)
Number analyzed (Participants) | 45 | 45 | 36 | 36
Number analyzed (Nights Analyzed) | 955 | 941 | 769 | 755
percentage of time | 6 [4 to 9] | 4 [3 to 8] | 6 [5 to 12] | 7 [4 to 10]
Statistical Analysis 1: Comparison: Pump Suspension Algorithm (Participants 11-14 Years) vs Standard of Care (Participants 11-14 Years); Test type: Superiority or Other; p = 0.18, t-test, 2 sided
Statistical Analysis 2: Comparison: Pump Suspension Algorithm (Participants 4-10 Years) vs Standard of Care (Participants 4-10 Years); Test type: Superiority or Other; p = 0.77, t-test, 2 sided

7. Secondary Outcome: Mean Morning Blood Glucose
Description: as for outcome 2
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Units Other Than Participants: Nights analyzed
Arm/Group | Pump Suspension Algorithm (Participants 11-14 Years) | Standard of Care (Participants 11-14 Years) | Pump Suspension Algorithm (Participants 4-10 Years) | Standard of Care (Participants 4-10 Years)
Number analyzed (Participants) | 45 | 45 | 36 | 36
Number analyzed (Nights analyzed) | 955 | 941 | 769 | 755
mg/dL | 176 (28) | 159 (29) | 158 (22) | 154 (25)
Statistical Analysis 1: Comparison: Pump Suspension Algorithm (Participants 11-14 Years) vs Standard of Care (Participants 11-14 Years); Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Pump Suspension Algorithm (Participants 4-10 Years) vs Standard of Care (Participants 4-10 Years); Test type: Superiority or Other; p = 0.11, t-test, 2 sided

8. Secondary Outcome: Percentage of Mornings With Blood Glucose >250 mg/dL (>13.9 mmol/L)
Description: as for outcome 2
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Population: as for outcome 2
Measure: Number; unit: percentage of mornings
Units Other Than Participants: Nights analyzed
Arm/Group | Pump Suspension Algorithm (Participants 11-14 Years) | Standard of Care (Participants 11-14 Years) | Pump Suspension Algorithm (Participants 4-10 Years) | Standard of Care (Participants 4-10 Years)
Number analyzed (Participants) | 45 | 45 | 36 | 36
Number analyzed (Nights analyzed) | 955 | 941 | 769 | 755
percentage of mornings | 11 | 10 | 7 | 9
Statistical Analysis 1: Comparison: Pump Suspension Algorithm (Participants 11-14 Years) vs Standard of Care (Participants 11-14 Years); Test type: Superiority or Other; p = 0.57, t-test, 2 sided
Statistical Analysis 2: Comparison: Pump Suspension Algorithm (Participants 4-10 Years) vs Standard of Care (Participants 4-10 Years); Test type: Superiority or Other; p = 0.18, t-test, 2 sided

9. Secondary Outcome: Morning Blood Ketones >=1.0 mmol/L
Description: as for outcome 2
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Population: as for outcome 2
Measure: Number; unit: percentage of mornings
Units Other Than Participants: Nights analyzed
Arm/Group | Pump Suspension Algorithm (Participants 11-14 Years) | Standard of Care (Participants 11-14 Years) | Pump Suspension Algorithm (Participants 4-10 Years) | Standard of Care (Participants 4-10 Years)
Number analyzed (Participants) | 45 | 45 | 36 | 36
Number analyzed (Nights analyzed) | 955 | 941 | 769 | 755
percentage of mornings | 1.0 | 0.4 | 2.3 | 2.9
Statistical Analysis 1: Comparison: Pump Suspension Algorithm (Participants 11-14 Years) vs Standard of Care (Participants 11-14 Years); Test type: Superiority or Other; p = 0.16, t-test, 2 sided
Statistical Analysis 2: Comparison: Pump Suspension Algorithm (Participants 4-10 Years) vs Standard of Care (Participants 4-10 Years); Test type: Superiority or Other; p = 0.39, t-test, 2 sided

10. Secondary Outcome: Percent of Mornings With Urine Ketones >/= 15 mg/dl
Description: Urine ketones measured each morning with Ketostix.
Time Frame: Overnight from system activation to deactivation in the morning upon awakening for 42 nights of system use
Population: as for outcome 2
Measure: Number; unit: percentage of mornings
Units Other Than Participants: Nights analyzed
Arm/Group | Pump Suspension Algorithm (Participants 11-14 Years) | Standard of Care (Participants 11-14 Years) | Pump Suspension Algorithm (Participants 4-10 Years) | Standard of Care (Participants 4-10 Years)
Number analyzed (Participants) | 45 | 45 | 36 | 36
Number analyzed (Nights analyzed) | 955 | 941 | 769 | 755
percentage of mornings | 1.7 | 1.4 | 3.5 | 2.6
Statistical Analysis 1: Comparison: Pump Suspension Algorithm (Participants 11-14 Years) vs Standard of Care (Participants 11-14 Years); Test type: Superiority or Other; p = 0.53, t-test, 2 sided
Statistical Analysis 2: Comparison: Pump Suspension Algorithm (Participants 4-10 Years) vs Standard of Care (Participants 4-10 Years); Test type: Superiority or Other; p = 0.28, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Study duration was about 3 months.
Arm/Group | Randomized Nights- Treatment or Control
Serious Adverse Events (participants affected / at risk) | 0/97
Other Adverse Events (participants affected / at risk) | 1/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Nights- Treatment or Control (N=97)
methicillin resistant Staphylococcus aureus (Infections and infestations) | 1 (1) — Infection at pump infusion set site.

LIMITATIONS AND CAVEATS:
Only selected participants prone to nocturnal hypoglycemia and only tested one continuous glucose sensor. Participants didn't know if system was active before activation so could not observe what would happen if the participants knew it was.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No